CLINICAL TRIAL: NCT04591275
Title: Randomized, Doubel-blinded, Parallel, Active-controlled Phase III Study, to Evaluate the Efficacy and Safety of CMAB807 Treatment Compared with Prolia® in Chinese Postmenopausal Women with Osteoporosis At High Risk of Fracture.
Brief Title: Clinical Efficacy and Safety Comparative Study Between CMAB807 Injection and Prolia® .
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Biomabs Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB807-III-001
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMAB807 (Experimental): 60mg, every 6 months, subcutaneously for twice. dietary supplement: elemental calcium orally, 600mg, daily, and vitamin D orally, 400IU, daily
  Interventions: Drug: CMAB807 Injection
- Prolia® (Active Comparator): 60mg, every 6 months, subcutaneously for twice. dietary supplement: elemental calcium orally, 600mg, daily, and vitamin D orally, 400IU, daily
  Interventions: Drug: Prolia®

INTERVENTIONS:
Drug: CMAB807 Injection — mAb targeting RANKL, human monoclonal antibody targeting RANKL
  Other Names: Denosumab Injection
  Arms: CMAB807
Drug: Prolia® — mAb targeting RANKL, human monoclonal antibody targeting RANKL
  Other Names: Denosumab Injection
  Arms: Prolia®

SUMMARY:
evaluate the differences in effectiveness and safety between CMAB807( potential biosimilar) and Prolia(original product)

DETAILED DESCRIPTION:
this is a randomized, double-blinded, parallel, active-controlled clinical phase III study. the primary objective is to evaluate the efficacy and safety of CMAB807 treatment compared with Prolia in Chinese postmenopausal women with osteoporosis at high risk of fracture.

Subjects should sequentially enrolled according to the protocol in one of two arms. Subjects who entered in test arm would receive 60mg of CMAB807 subcutaneously every 6 months for one year, while those who entered in control arm should receive 60mg of Prolia subcutaneously every 6 months for one year. Meanwhile, every subject should taking 600mg calcium and 400IU vitamin D daily from successfully screening to the end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed, understood, voluntary participate, and the patient himself or guardian agree to sign the written informed consent and patient be able to comply with the protocol;
2. Aged from 50 years to 85 years, inclusive;
3. Spontaneous amenorrhea time ≥ 2 years, or bilateral oophorectomy≥ 2 years. If the status of bilateral ovariectomies is unknown, the menopause status should be confirmed by follicle stimulating hormone(FSH) level≥ 40IU/L;
4. Based on the results of dual energy X-ray absorptiometry, BMD of lumbar spine(L1~L4), femoral neck or total hip: -4.0<T-Score≤-2.5；
5. There must be at least one of the following risk factors:

   * History of osteoporotic fracture;
   * Father's and mother's hip fracture history, or both parents';
   * Low body mass index(≤19kg/m^2);
   * Patient's age was equal or greater than 70 years old;
   * Current smoker;
   * CTX1 was one standard deviation higher than that of healthy premenopausal women within screening period(ie, CTX1>0.43ng/mL);
6. Ability to act independently.

Exclusion Criteria:

1. Suffering from the following diseases known to affect calcium or bone metabolism:

   * Various metabolic bone diseases, such as osteogenesis imperfecta and osteomalacia;
   * Paget's osteopathy;
   * Cushing's syndrome;
   * Hyperprolactinemia;
   * Hypopituitarism;
   * Acromegaly;
   * History of hyperparathyroidism or hypoparathyroidism;
   * History of hyperthyroidism or hypothyroidism(hypothyroidism patients can be included: only receiving stable thyroid hormone replacement therapy, if the thyroid stimulating hormone(TSH) level is normal, or 5.5μIU/mL<TSH≤10.0μIU/mL, and free thyroxine(FT4) is in normal range can be included);
   * Malabsorption syndrome or various gastrointestinal diseases associated with malabsorption, such as Crohn's disease and chronic pancreatitis;
   * Abnormal level of blood calcium: the current diagnosis of hypocalcemia or hypercalcemia or albumin corrected serum calcium levels are not within the laboratory normal range(calcium supplements should not be used for at least 8 hours prior to serum calcium testing);
   * Vitamin D deficiency: 25 hydroxyvitamin D concentration<20ng/mL. Allowed to retest after oral vitamin D2 soft capsules in the screening period. If the concentration of 25 hydroxyvitamin D is more than or equal to 20ng/mL， it can be selected;
   * Other diseases such as rheumatoid arthritis, gout, multiple myeloma, etc;
2. Medical history of two or more vertebrae fractures;
3. Malignant tumor(excluding skin basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ or breast ductal carcinoma in situ) in recent 5 years;
4. Severe renal function damage(creatinine clearance rate<30mL/min), or dialysis, urinary calculi or chronic cystitis;
5. Suffering from the following liver or biliary diseases:

   * Liver cirrhosis;
   * Biliary abnormalities(except for Gilbert syndrome or asymptomatic gallstones);
   * Positive hepatitis C virus antibody(HCV-Ab) and the titer of HCV-RNA exceeded the upper limit of norma;
   * Positive hepatitis B suface antigen(HBsAg) and peripheral blood HBV-DNA titer ≥1000 capies[CPS]/mL or 200IU/mL;
   * Unstable liver disease: defined as liver ascites, hepatic encephalopathy, coagulopathy, hypoalbuminemia, varicosis in esophagus or stomach fundus or persistent hepatic jaundice;
6. Liver transaminase: aspartate aminotransferase≥2.0×upper limit of norma value(ULN), alanine aminotransferase≥2.0ULN, alkaline phosphatase≥1.5ULN or total bilirubin≥1.5ULN;
7. Suffering from the following oral diseases:

   * Osteomyelitis or osteonecrosis of the jaw, previously or currently;
   * Actue dental or mandibular disease requiring stomatological surgery;
   * Planned invasive dental surgery during the trial period;
   * Dental or stomatological surgery have not healed;
8. Conditions which can influence bone mineral density determination by dual energy X-ray absorptiometry:

   * Less than two lumbar vertebrae can be measured;
   * Height, weight or waistline may hinder accurate measurement;
   * Other conditions that may affect bone density testing
9. Received anti-osteoporosis drugs or those drugs may affect bone metabolism:

   * Use of injectable bisphosphonates, fluoride or strontium within 2 years before screening;
   * Use of oral bisphosphonates: more than 2 years, or more than 3 months but less than 2 years and discontinued from last dosage less than 1 year, simultaneously;
   * Usage of any drugs which may affect bone metabolism within 6 weeks before screening: parathyroid hormone or parathyroid hormone analogue(such as teriparatide); assimilative hormone or testosterone; glucocorticoid(equivalent to prednisone>5mg/day for more than 10 days); systemic hormone replacement therapy; selective estrogen receptor regulator(such as reloxifene); tibolone; calcitonin; active vitamin D and ite analogues, other bone active drugs include anticonvulsant drugs(except benzodiazepines) and he[arin; long-term systemic use of ketoconazole, androgen, adrenocorticotropic hormone, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, gonadotropin releasing hormone agonist;
   * Patients who have received RANKL inhibitors previously;
10. Positive HIV antibody;
11. Known alcoholism or drug abuse(during 12 months before screening), because alcohol or drug abuse may interfere with subject's understanding or finish of trial;
12. Known allergy to test drug, reference drug or basic drug and its excipients;
13. Participate in interventionary clinical study(drug or device) within one month before screening;
14. Other serious, acute or chronic diseases, mental disorders or laboratory abnormalities, which are judged by investigator to be unsuitable to participate this study.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
BMD percentage change from baseline at lumbar spine(L1~L4) | baseline, at 12 months
  Percentage change from baseline at lumbar spine(L1~L4) by dual-energy X-ray absorptiometry to month 12 of treatment and compare between two arms. Percentage change of lumbar spine BMD from baseline to at month 12 of treatment=(BMD at month 12 of treatment - BMD at baseline)/BMD at baseline*100%

SECONDARY OUTCOMES:
BMD percentage change from baseline at lumbar spine(L1~L4) | baseline, at 6 months
  Percentage change from baseline at lumbar spine(L1~L4) by dual-energy X-ray absorptiometry to month 6 of treatment and compare between two arms. Percentage change of lumbar spine BMD from baseline to at month 12 of treatment=(BMD at month 12 of treatment - BMD at baseline)/BMD at baseline*100%
BMD percentage change from baseline at total hip, trochanter and femoral neck | baseline, at month 6, at month 12
  Pencentage change from baseline at total hip, trochanter and fremoral neck by dual-energy-X-ray absorptiometry to month 6 and month 12 of treatment, and compare between two arms. Percentage to total hip, trochanter and femoral neck BMD from baseline at month 6 or month 12 of treatment=(BMD at month 6 or month 12 of treatment - BMD at baseline)/BMD at baseline*100%
Serum CTX1 and P1NP concentration percentage change from baseline | baseline, at month 1, at month 3, at month 6, at month 9,and at month 12
  Fasting serum CTX1 and P1NP samples should be collected. Percentage changes of serum CTX1 or P1NP concentrations from baseline at month 1, month 3, month 6, month 9 and at month 12 of treatment=(serum concentrations at month 1, month 3, month 6, month 9 and month 12 - serum concentration at baseline)/serum concentration at baseline*100%
Proporation of new osteoporotic fractures(vertebrae, total hip and non-vertebrae) occurring within the study period | baseline, at month 12
  Osteoporotic fracture is defined as the fracture occurred when subject suffers minor trauma or during daily activities. Common occurrence sites are vertebral body, hip, distal forearm, proximal humerus and pelvis, etc
Adeverse events and serious adverse events | baseline ,at 12 months
  Evaluation of the drug reactions, changes in physical examination findings, changes in vital signs, stomatological examination, clinical laboratory testing for systemic safety(including complete blood count, urinalysis, clinical chemistries, coagulation function, liver function, renal function, parathyroid function), and electrocardiography
Immunogenicity | baseline, at 12 months
  Binding antibody and neutralizing antibody formation assays were used to assess number of subjects with anti-denosumab antibody
Population pharmacokinetics analysis | baseline, at 12 months
  The pharmacokinetic parameters were described statistically, such as population typical value of clearance rate, estimation precision of typical value, confindence interval of typical value, and inter individual variation

CONTACTS AND LOCATIONS:
Overall Officials: weibo Xia, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No